CLINICAL TRIAL: NCT00547456
Title: Consequences of Nocturnal and Daytime Hypoxemia in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 05.02.097
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decrease in oxygen level when sleeping (Other): Patients are their own controls and tested pre and post the addition of night time supplemental oxygen
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Oxygen 2-3L Nasal cannula

SUMMARY:
We will determine whether oxygen therapy lowers the level of substances in the blood which cause inflammation, which is one of the adverse effects of COPD and whether oxygen improves overall well being and quality of life as well as sleep quality.

DETAILED DESCRIPTION:
Hypothesis: Isolated nocturnal hypoxemia contributes to chronic systemic inflammation in COPD by activating circulating neutrophils.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females with a diagnosis of COPD screened for nocturnal desaturation as indicated above.
* Clinical stability defined by absence of treatment change or need for acute care within the last two months.
* Weight stable, within 5%, in the previous three months as measured during office visits.
* Willingness to participate in a clinical study.

Exclusion Criteria:

* Acute illness within the preceding 2 months.
* Patients who received systemic glucocorticoid therapy within the past month.
* Clinical and/or overnight pulse oximetry evidence of obstructive sleep apnea (OSA). The Multivariate Apnea Prediction Questionnaire (MAP) will be given to all patients to assess the likelihood of OSA based on common symptoms of this disorder. While we recognize that this screening instrument was not evaluated specifically in COPD patients, it assesses common signs and symptoms of OSA. This tool has been shown to identify OSA with 95% sensitivity (63). In addition, the ODI 4% will be determined from the overnight pulse oximetry recording. Patients will be excluded if the MAP score is > 0.4 or if the ODI 4% is >15/hour, which is suggestive of the concomitant presence of obstructive sleep apnea.
* Hypercapnia defined as PaCO2 > 50 mmHg on resting arterial blood gas
* Previous diagnosis of erythrocytosis, pulmonary vascular disease, pleural effusions, ischemic heart disease or congestive heart failure.
* No chronic illnesses known to affect the inflammatory response such as infection, collagen vascular disease, liver disease, thyroid disease or diabetes.
* Primary care or pulmonary physician refusal.
* Patient refusal for any reason.
* Lack of capacity to participate in the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Cohen, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore LIJ Health System, New Hyde Park, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment details occurred as outlined in protocol
Period: Overall Study
Arm/Group | Decrease in Oxygen Level When Sleeping
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decrease in Oxygen Level When Sleeping
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — participants between the ages of 18-65
  Participants
    <=18 years | 0
    Between 18 and 65 years | 20
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [40 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20
nocturnal hypoxemia [Number; unit: participants] | 20
Number of Participants with Nocturnal and Daytime Hypoxemia in COPD [Number; unit: participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Demonstration of Improvement in Systemic Inflammation, Sleep Quality and Health Related Quality of Life With Nocturnal Oxygen Supplementation.
Time Frame: 4 weeks
Population: The assay used did not work, as a result, no data for any Outcome Measures was collected. The trial is closed and completed.
Arm/Group | Decrease in Oxygen Level When Sleeping
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Decrease in Oxygen Level When Sleeping
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes